CLINICAL TRIAL: NCT05392868
Title: A Clinical Protocol on the Effectiveness of 38% Silver Diamine Fluoride in Reducing Dentine Hypersensitivity on Exposed Root Surface in Older Chinese Adults
Brief Title: Managing Dentine Hypersensitivity With Silver Diamine Fluoride on Older Adults
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chun Hung Chu, Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HKU2022
Record Dates: First submitted 2022-05-22; First posted 2022-05-26 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Dentine Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SDF (Experimental): 38% silver diamine fluoride solution
  Interventions: Device: SDF
- KNO3 (Active Comparator): 5% potassium nitrate solution
  Interventions: Device: KNO3

INTERVENTIONS:
Device: SDF — 38% silver diamine fluoride solution
  Arms: SDF
Device: KNO3 — 5% potassium nitrate solution
  Arms: KNO3

SUMMARY:
Background: Dentine hypersensitivity is a common oral complaint from older adults. It induces pain, affects oral hygiene practice, limits food choices and negatively affects the quality of life. Silver diamine fluoride (SDF) is a desensitizing agent but well-designed clinical trials are lacking. The objective of this study is to evaluate the effectiveness of SDF in reducing dentine hypersensitivity in older Chinese adults.

Methods: This is a double-blinded randomised clinical trial recruiting 166 healthy older adults aged 65 or over after having written consent. A trained calibrated examiner will conduct clinical examination and assess dentine hypersensitive using a blast of compressed air delivered from 3-in-1 syringe. Older adults with a tooth with a self-perceived sensitivity score (SS) of 8 or above will be recruited. They will then be block randomised to receive either 38% SDF solution or 5% potassium nitrate every 4 weeks on the exposed root surface of the most hypersensitive tooth. The visible plaque index, bleeding on probing and probing depth (mm) will be recorded on the most hypersensitive tooth. The same examiner will perform clinical examination and assess the dentine hypersensitivity using the same tools and methods at 4-week and 8-week follow-ups. The examiner and older adults will be blinded to treatment allocation. The primary outcome is the percentage of change in SS before and after intervention at 8 weeks. The secondary outcome will be the percentage of change in VPI before and after intervention at 8 weeks.

Clinical significance: It will provide evidence to manage dentine hypersensitivity in older adults in clinical care.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy;
* no known or suspected allergy to the study ingredients or materials
* have all active dental diseases under control but reported hypersensitivity

Exclusion Criteria:

* using any desensitizing agent within one month
* have major systemic diseases such as cancer
* receive medications that may affect pain perception within one month
* have dentine hypersensitivity due to other dental conditions such as caries
* are not able to give written consent

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in dentine hypersensitivity | at 8-week follow-up
  the percentage of change in self-perceived sensitivity score (SS)

SECONDARY OUTCOMES:
Change in oral hygiene status | at 8-week follow-up
  the percentage of change in visible plaque index

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan AKY, Tsang YC, Jiang CM, Leung KCM, Lo ECM, Chu CH. Treating hypersensitivity in older adults with silver diamine fluoride: A randomised clinical trial. J Dent. 2023 Sep;136:104616. doi: 10.1016/j.jdent.2023.104616. Epub 2023 Jul 14. PMID 37454789
- [Derived] Chan AKY, Tamrakar M, Jiang CM, Tsang YC, Leung KCM, Chu CH. Effectiveness of 38% Silver Diamine Fluoride in Reducing Dentine Hypersensitivity on Exposed Root Surface in Older Chinese Adults: Study Protocol for a Randomised Double-Blind Study. Dent J (Basel). 2022 Oct 19;10(10):194. doi: 10.3390/dj10100194. PMID 36286004